CLINICAL TRIAL: NCT00179621
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, 3-Arm Study of the Efficacy and Safety of 2 Doses of Lenalidomide Versus Placebo in Red Blood Cell (RBC) Transfusion-Dependent Subjects With Low- or Intermediate-1-Risk Myelodysplastic Syndromes Associated With a Deletion (Del) 5q[31] Cytogenetic Abnormality
Brief Title: Lenalidomide Versus Placebo in Myelodysplastic Syndromes With a Deletion 5q[31] Abnormality
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Jay Backstrom, MD, Vice President, Clinical Development MDS, Celgene Corporation
Organization: Celgene (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-5013-MDS-004; 2005-000454-73 (EudraCT Number)
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Results first posted 2011-03-17 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS; transfusion dependent; anaemia; cytogenetic abnormality 5q-; erythroid response; leukaemia; CC-5013; Celgene; revlimid; lenalidomide
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia; Leukemia | interventions — Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo matching to active study arms.
  Interventions: Drug: Placebo
- Lenalidomide 5 mg (Experimental): Lenalidomide 5 mg daily 28/28 days
  Interventions: Drug: Lenalidomide 5 mg
- Lenalidomide 10 mg (Experimental): Lenalidomide 10 mg daily 21/28 days
  Interventions: Drug: Lenalidomide 10 mg

INTERVENTIONS:
Drug: Lenalidomide 5 mg — Lenalidomide 5 mg daily 28/28 days
  Other Names: Revlimid
  Arms: Lenalidomide 5 mg
Drug: Lenalidomide 10 mg — Lenalidomide 10 mg daily 21/28 days
  Other Names: Revlimid
  Arms: Lenalidomide 10 mg
Drug: Placebo — Placebo, matching to active study drug arms
  Arms: Placebo

SUMMARY:
The purpose of this study was to compare 2 doses (10 mg and 5 mg) of lenalidomide to that of placebo in subjects with red blood cell (RBC) transfusion-dependent low- or intermediate-1-risk IPSS MDS associated with a deletion (del) 5q[31] cytogenetic abnormality. Study participants were randomized to one of the two treatment groups or to placebo and took the study drug for 16 weeks. At this timepoint, participants were evaluated for erythroid response. If participants did not achieve at least a minor erythroid response, they were discontinued from the Double-Blind phase and entered into the Open-Label phase. All erythroid responders at Week 16 were to continue in the Double-Blind phase for up to 52 weeks. For participants that were still responding at the end of Double-Blind phase, they could then rollover into the Open-Label phase for an additional two years. Participants could remain on study for up to a total of 3 years. All participants who discontinued from the study were followed every 4 months for overall survival and progression to acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
MDS-004 was a multicenter, randomized, double-blind, placebo-controlled, 3-arm study of 2 doses of lenalidomide versus placebo administered to RBC transfusion-dependent adults with low- or intermediate-1 risk MDS associated with a del 5q[31] cytogentetic abnormality. Potential participants that had a del 5q[31] cytogenetic abnormality plus other additional cytogenetic abnormalities were also eligible for enrollment. Transfusion-dependent anemia was defined as documentation that a participant with anemia due to MDS did not have any consecutive 56 days (8 weeks) that were RBC transfusion free during at least the 112 days (16 weeks) prior to Day 1 of the Pre-Randomization Phase.

This study was conducted in three phases:

1. a Pre-Randomization Phase
2. a Double-Blind Treatment Phase
3. an Open-Label Extension Phase

Potentially protocol-eligible participants entered the Pre-Randomization Phase and were evaluated for the inclusion and exclusion criteria for the Double-Blind Treatment Phase. The Pre-Randomization Phase was not to last for more than 56 days (8 weeks). When the participant's baseline RBC transfusion requirement was calculated, and it had been determined that all eligibility criteria had been met, the participant could be randomized for treatment in the Double-Blind Treatment Phase at the time of their next RBC transfusion. This RBC transfusion had to occur within 56 days of the participant's last previous RBC transfusion.

Participants meeting eligibility criteria were randomized (1:1:1 ratio) to receive either lenalidomide 10 mg/day on days 1-21, lenalidomide 5 mg/day on days 1-28, or placebo on days 1-28; all on a 28-day cycle. Randomization was performed using a validated interactive voice response system. Participants were stratified according to karyotype (IPSS karyotype score: 0 vs > 0; i.e., isolated del 5q[31] vs del 5q[31] plus ≥ 1 additional cytogenetic abnormality). A complete blood count (CBC), serum or plasma ferritin, and EPO levels were measured to determine baseline levels.

Participants who achieved at least a minor erythroid response (i.e. 50% decrease in transfusion requirements) by week 16 could continue treatment in the Double-Blind phase for up to 52 weeks, unless there was evidence of erythroid relapse, disease progression, or unacceptable toxicity. Those who did not achieve at least a minor erythroid response by week 16 were discontinued from the Double-Blind phase for lack of therapeutic efficacy, and unblinded and were potentially eligible for Open-Label treatment. All participants who completed the double-blind treatment phase (the first 52 weeks of the trial) without disease progression or erythroid relapse were unblinded and entered the Open-Label extension phase at their current lenalidomide dose. Participants in the placebo or lenalidomide 5 mg arms who failed to achieve at least a minor erythroid response by week 16 or who had an erythroid relapse could cross over to lenalidomide 5 mg or 10 mg, respectively, in the Open-Label Extension phase.

Lenalidomide treatment could be continued in the Open-label Extension phase for up to 3 years (156 weeks) of total study participation. Participants with disease progression at any time and participants in the lenalidomide 10 mg group who did not achieve at least a minor erythroid response by week 16 were withdrawn from the study and were ineligible for Open-Label treatment.

Serial measurements for efficacy and safety were performed every 28 days. In addition, CBCs were monitored weekly for the first 8 weeks, every 2 weeks for the next 8 weeks, and every 4 weeks thereafter. Bone marrow aspirate (BMA) and standard cytogenetic studies were performed at baseline, weeks 12, week 24, and every 24 weeks thereafter and when clinically indicated for assessment of disease progression. BMAs were submitted for central pathology review and sent to a central cytogenetics laboratory for processing and review. All participants were followed for overall survival (OS) and progression to acute myeloid leukemia (AML).

Lenalidomide or placebo dosing was reduced for dose-limiting toxicities according to the following dose reduction schedule:

* Lenalidomide 5 mg (starting dose)

  * dose level -1 (5 mg every other day)
  * dose level -2 (5 mg twice a week)
  * dose level -3 (5 mg weekly)
* Lenalidomide 10 mg (starting dose)

  * dose level -1 (5 mg daily)
  * dose level -2 (5 mg every other day)
  * dose level -3 (5 mg twice a week)

Participants who could not tolerate dose level -3 discontinued treatment. For grade 4 neutropenia, lenalidomide was required per protocol to be interrupted and resumed at a decreased dose level when the absolute neutrophil count (ANC) recovered to ≥ 500/μL. For grade 4 thrombocytopenia, lenalidomide was interrupted and then resumed at a decreased dose level when the platelet count recovered to: between ≥ 25,000/μL and < 50,000/μL on at least 2 occasions for ≥ 7 days; or ≥ 50,000 at any time, respectively. Prophylactic and therapeutic use of granulocyte colony-stimulating factors (G-CSF) or granulocyte macrophage colony-stimulating factors (GM-CSF) was allowed.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form
* Age 18 years at the time of signing the informed consent form
* Documented diagnosis of myelodysplastic syndromes (MDS) that meets International Prognostic Scoring System (IPSS) criteria for low to intermediate-1-risk disease and has an associated del 5q(31) cytogenetic abnormality
* Red blood cell (RBC) transfusion dependent anaemia defined as not having any 56 days without a RBC transfusion within at least the immediate 112 days
* Must be able to adhere to the study visit schedule and other protocol requirements
* Women of childbearing potential must have a negative pregnancy test prior to inclusion

Exclusion Criteria:

* Pregnant or lactating females
* Prior therapy with lenalidomide
* Proliferative (white blood cell (WBC)= 12,000/mL) chronic myelomonocytic leukemia (CMML)
* Prior >= grade-2 (using the National Cancer Institute (NCI)'s Common Terminology Criteria for AEs (CTCAE) (v 3.0)) allergic reaction to thalidomide
* Prior desquamating (blistering) rash while taking thalidomide
* Prior history of malignancy other than MDS (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been free of disease for >3 years
* Use of cytotoxic chemotherapeutic agents or experimental agents (agents that are not commercially available) for the treatment of MDS within 28 days
* Less than 6 months since prior allogeneic bone marrow transplantation
* Less than 3 months since prior autologous bone marrow or stem cell transplantation
* Less than 28 days since prior myelosuppressive anticancer biologic therapy
* Recombinant human erythropoietin (rHuEPO) therapy received within 28 days
* Known human immunodeficiency virus (HIV-1) positivity
* Any serious medical condition or psychiatric illness that will prevent the subject from signing the informed consent form or will place the subject at unacceptable risk if he or she participates in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2005-07; Primary Completion 2008-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Backstrom, MD, Study Director — Celgene Corporation
Locations (38):
- Belgium (4):
  - AZ St-Jan Brugge AV, Bruges
  - UZ Gent, Ghent
  - UZ Gasthuisberg, Leuven
  - CHU Mont Godine, Yvoir
- France (12):
  - Institut Paoli-Calmettes, Marseille, Cedex 9
  - CHU d'Angers Service des Maladies du Sang, Angers
  - Hopital Avicenne, Bobigny
  - CHRU Lille Service des Maladies du Sang, Lille
  - CHU Nantes Hematologie et Medicine interne, Nantes
  - CHU Archet 1Hematologie Clinique, Nice
  - Hôpital Cochin Hematologie Clinique, Paris
  - Centre Jean Bernhard Service Onco-Hematologie, Poitiers
  - Centre Henri Becquerel Service d'Hematologie Clinique, Rouen
  - CHU Purpan, Place du Dr Baylac, Pavillon des Médecines, Toulouse
  - CHU Purpan, Place du Dr. Baylac, Pavillion des Medecines, Toulouse
  - CHU Nancy Hematologie et Medecine interne, Vandœuvre-lès-Nancy
- Germany (4):
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - St Johannes Hospital, Duisburg
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Hannover Medical School, Hanover
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (2):
  - Ospedale Niguarda Ca Granda, Milan
  - University of Pavia Division of Hematology, Pavia
- Netherlands (2):
  - University of Medical Centre, Nijmegen
  - Hematologie Erasmus MC, Rotterdam
- Spain (2):
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario La Fe, Valencia
- Sweden (3):
  - SU/Sahlgrenska Section of Hematology & Coagulation, Gothenburg
  - Department of Medicine University Hospital, Lund
  - Korolinska Institutet Department of Hematology, Stockholm
- United Kingdom (8):
  - University Hospital of Wales, Dept of Haematology, Cardiff, Wales
  - Leed General Infirmary, Leeds, West Yorkshire
  - The Royal Bournemouth Hospital, Bournemouth
  - Ninewells Hospital and Medical School, Dundee
  - Kings College Hospital, Denmark Hill, London
  - Central Manchester and Manchester Children's University Hospitals NHS Trust, Manchester
  - Nottingham City Hospital, Nottingham
  - John Radcliffe Hospital and the Weatherall Institute of Molecular Medicine, Oxford

REFERENCES:
- [Result] Fenaux, Pierre, Giagounidis, Aristotle, Selleslag, Dominik, Beyne-Rauzy, Odile, Mufti, Ghulam J, Mittelman, Moshe, Muus, Petra, te Boekhorst, Peter, Sanz, Guillermo, del Canizo, Consuelo, Guerci-Bresler, Agnes, Schlegelberger, Brigitte, Aul, Carlo, Kreipe, Hans, Goehring, Gudrun, Knight, Robert, Francis, John, Fu, Tommy, Hellstrom-Lindberg, Eva. RBC Transfusion Independence and Safety Profile of Lenalidomide 5 or 10 mg in Pts with Low- or Int-1-Risk MDS with Del5q: Results From a Randomized Phase III Trial (MDS-004). ASH Annual Meeting Abstracts 2009 114: 944.
- [Result] Fenaux, P., Giagounidis, A., Selleslag, D. L., Beyne-Rauzy, O., Mittelman, M., Muus, P., Knight, R. D., Fu, T., Hellstrom-Lindberg, E., The MDS-004 Len del(5q) Study Group. Safety of lenalidomide (LEN) from a randomized phase III trial (MDS-004) in low-/int-1-risk myelodysplastic syndromes (MDS) with a del(5q) abnormality. J Clin Oncol (Meeting Abstracts) 2010 28: 6598
- [Result] Fenaux, P., Giagounidis, A., Selleslag, D., Knight, R., Fu, T., Hellström-Lindberg, E. Effect of baseline EPO and prior erythropoiesis stimulating agents on RBC transfusion independence in Low-/Int-1-Risk MDS with del 5q treated with lenalidomide: A randomized phase 3 study (MDS-004). Haematologica 2010; 95[suppl.2]:125, abs. 0311.
- [Result] Brandenburg, N., Fu, T., Revicki, D., Knight, R., Muus, P., Fenaux, P. Impact of lenalidomide on health-related quality of life in patients with RBC transfusion-dependent low- or int-1-risk myelodysplastic syndromes with del 5q: a randomized Phase 3 study (MDS-004). Haematologica 2010; 95[suppl.2]:127, abs. 0316
- [Result] Fenaux, P., Giagounidis, A., Beyne-Rauzy, O., Mufti, G., Mittelman, M., Muus, P., te Boekhorst, P., Sanz, G., Cazzola, M., Backstrom, J., Fu, T., Hellström-Lindberg, E. Prognostic Factors of Long-Term Outcomes In Low- or Int-1-Risk MDS with del5q Treated with Lenalidomide (LEN): Results From a Randomized Phase 3 Trial (MDS-004). Blood ASH Annual Meeting Abstracts 2010 116:21 abs. 4027.
- [Result] Brandenburg, N., Yu, R., Revicki, D. Reliability and Validity of the FACT-AN In Patients with Low or Int-1-Risk Myelodysplastic Syndromes with Deletion 5q. Blood ASH Annual Meeting Abstracts 2010 116:21 abs. 3827.
- [Derived] Fenaux P, Giagounidis A, Selleslag D, Beyne-Rauzy O, Mittelman M, Muus P, Nimer SD, Hellstrom-Lindberg E, Powell BL, Guerci-Bresler A, Sekeres MA, Deeg HJ, Del Canizo C, Greenberg PL, Shammo JM, Skikne B, Yu X, List AF. Clinical characteristics and outcomes according to age in lenalidomide-treated patients with RBC transfusion-dependent lower-risk MDS and del(5q). J Hematol Oncol. 2017 Jun 26;10(1):131. doi: 10.1186/s13045-017-0491-2. PMID 28651604
- [Derived] Saft L, Karimi M, Ghaderi M, Matolcsy A, Mufti GJ, Kulasekararaj A, Gohring G, Giagounidis A, Selleslag D, Muus P, Sanz G, Mittelman M, Bowen D, Porwit A, Fu T, Backstrom J, Fenaux P, MacBeth KJ, Hellstrom-Lindberg E. p53 protein expression independently predicts outcome in patients with lower-risk myelodysplastic syndromes with del(5q). Haematologica. 2014 Jun;99(6):1041-9. doi: 10.3324/haematol.2013.098103. Epub 2014 Mar 28. PMID 24682512
- [Derived] Fenaux P, Giagounidis A, Selleslag D, Beyne-Rauzy O, Mufti G, Mittelman M, Muus P, Te Boekhorst P, Sanz G, Del Canizo C, Guerci-Bresler A, Nilsson L, Platzbecker U, Lubbert M, Quesnel B, Cazzola M, Ganser A, Bowen D, Schlegelberger B, Aul C, Knight R, Francis J, Fu T, Hellstrom-Lindberg E; MDS-004 Lenalidomide del5q Study Group. A randomized phase 3 study of lenalidomide versus placebo in RBC transfusion-dependent patients with Low-/Intermediate-1-risk myelodysplastic syndromes with del5q. Blood. 2011 Oct 6;118(14):3765-76. doi: 10.1182/blood-2011-01-330126. Epub 2011 Jul 13. PMID 21753188
- [Derived] Gohring G, Giagounidis A, Busche G, Hofmann W, Kreipe HH, Fenaux P, Hellstrom-Lindberg E, Schlegelberger B. Cytogenetic follow-up by karyotyping and fluorescence in situ hybridization: implications for monitoring patients with myelodysplastic syndrome and deletion 5q treated with lenalidomide. Haematologica. 2011 Feb;96(2):319-22. doi: 10.3324/haematol.2010.026658. Epub 2010 Nov 25. PMID 21109690

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 263 potential participants were screened. Potentially protocol-eligible participants were then entered into the Pre-Randomization Phase (up to 56 days) to ensure eligibility criteria were met prior to entering the Double-Blind Phase. A total of 205 participants were randomized into the study.
Groups:
- Lenalidomide 5 mg: Lenalidomide 5 mg daily for 28 days
- Lenalidomide 10 mg: Lenalidomide 10 mg daily for 21 of 28 days
- Placebo Crossover to 5 mg Open-label Period: Participants receiving placebo in the Double-Blind phase and Lenalidomide in the Open-Label phase.
Period: Double-Blind Period
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg | Placebo Crossover to 5 mg Open-label Period
Started | 67 | 69 | 69 | 0
Completed | 3 | 23 | 39 | 0
Not Completed | 64 | 46 | 30 | 0
Not completed — Lack of Therapeutic Effect | 59 | 35 | 19 | 0
Not completed — Adverse Event | 2 | 7 | 4 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 0
Not completed — Death | 0 | 1 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Other | 0 | 2 | 2 | 0
Period: Open-Label Period
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg | Placebo Crossover to 5 mg Open-label Period
Started | 0 | 42 ('Started' includes 23 participants who completed double-blind and 19 who discontinued double-blind.) | 47 ('Started' includes 39 participants who completed double-blind and 8 who discontinued double-blind.) | 56 ('Started' includes 1 participant who completed double-blind and 55 who discontinued double-blind.)
Completed | 0 | 14 | 19 | 13
Not Completed | 0 | 28 | 28 | 43
Not completed — Lack of Therapeutic Effect | 0 | 19 | 19 | 31
Not completed — Adverse Event | 0 | 6 | 5 | 6
Not completed — Withdrawal by Subject | 0 | 2 | 2 | 2
Not completed — Death | 0 | 0 | 1 | 2
Not completed — Other | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg | Total
Number analyzed (Participants) | 67 | 69 | 69 | 205
Age Continuous [Median (Full Range); unit: years] | 69.9 [39.0 to 85.0] | 66.0 [40.0 to 86.0] | 68.0 [36.0 to 84.0] | 68.0 [36.0 to 86.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 53 | 49 | 156
  Male | 13 | 16 | 20 | 49
Race/Ethnicity, Customized [Number; unit: participants]
  White | 66 | 67 | 69 | 202
  Other | 1 | 2 | 0 | 3
5q- (31-33) Chromosomal Abnormality [Number; unit: Participants]
  Yes | 63 | 64 | 64 | 191
  No | 1 | 2 | 1 | 4
  Missing | 3 | 3 | 4 | 10
International Prognostic Scoring System (IPSS) [Number; unit: participants] — The international prognostic scoring system (IPSS) is a standard for risk assessment in primary myelodysplastic syndromes (MDS) that categorizes prognoses taking into account cytogenetics, cytopenias, blasts and blood counts. The IPSS prognostic subgroups consist of low-, intermediate-1-, intermediate-2-, and high-risk groups. The scale is 0-3.5 at 0.5 increments. Scores of 0=Low; 0.5-1.0=Int-1; 1.5-2.0=Int-2; 2.5-3.5=High risk which corresponds to poorer prognosis. The assessment was performed by the Central Reviewer.
  participants
    Low risk (0) | 30 | 20 | 20 | 70
    Intermediate-1 (0.5 - 1.0) | 22 | 29 | 23 | 74
    Intermediate-2 (1.5 - 2.0) | 2 | 5 | 3 | 10
    High Risk (≥ 2.5) | 0 | 0 | 1 | 1
    Missing data | 13 | 15 | 22 | 50
French-American-British (FAB) Classification [Number; unit: participants] — FAB is a classification system for five (5) subtypes of myelodysplastic syndrome that are distinguished by the percentage of myeloblasts, presence or absence of ringed sideroblasts or a monocytosis. Classification was made by the Central Reviewer.
  participants
    Refractory anemia (RA) | 37 | 38 | 32 | 107
    Refractory anemia with ringed sideroblasts (RARS) | 8 | 7 | 9 | 24
    Refractory anemia with excess blasts (RAEB) | 4 | 9 | 9 | 22
    Chronic myelomonocytic leukemia (CMML) | 1 | 2 | 0 | 3
    RAEB in transformation | 1 | 0 | 0 | 1
    Chronic myelogenous leukemia (CML) | 0 | 0 | 1 | 1
    Specimen not adequate from diagnosis | 12 | 11 | 17 | 40
    Other or missing | 4 | 2 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Achieved Red Blood Cell (RBC) Transfusion Independence for >= 26 Weeks (182 Days)
Description: The count of study participants who had no RBC transfusions for 26 consecutive weeks or more during the double-blind period.
Time Frame: Up to 52 weeks
Population: The modified intent-to-treat (mITT) population included all participants with centrally-confirmed Low- or Int-1-risk MDS with del 5q[31] and documented RBC transfusion dependence who had received ≥ 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg
Number analyzed (Participants) | 51 | 47 | 41
Participants | 3 | 20 | 23
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide 5 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — To compare the response rates of Lenalidomide 5 mg QD vs. placebo, the Hochberg procedure was used to control the familywise error rate of 0.05; Stratified by International Prognostic Scoring System (IPSS) score (IPSS combined score =0 versus >0) to compare lenalidomide treatment with placebo
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide 10 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — To compare the response rates of Lenalidomide 10 mg QD vs. placebo, the Hochberg procedure was used to control the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Participants Who Achieved Red Blood Cell (RBC) Transfusion Independence for 56 Days
Description: Count of study participants who had no RBC transfusions during any 56 or more consecutive study days during the double-blind period.
Time Frame: Up to 52 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg
Number analyzed (Participants) | 51 | 47 | 41
Participants | 4 | 24 | 25
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide 5 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide 10 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Duration of Red Blood Cell (RBC) Transfusion Independence for Participants Who Became RBC Transfusion Independent for at Least 182 Days
Description: Mean number of weeks that participants who achieved RBC transfusion independence for at least 182 days were able to maintain RBC transfusion independence. Both double-blind and open-label periods are included.
Time Frame: up to 3 years
Population: The modified intent-to-treat (mITT) population included all participants who achieved RBC transfusion independence for at least 182 days.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg
Number analyzed (Participants) | 3 | 20 | 23
Weeks | 61.4 (10.93) | 107.7 (52.35) | 108.6 (40.63)

4. Secondary Outcome: Maximum Change From Baseline in Hemoglobin During the Double-blind Period for Participants Who Became Red Blood Cell (RBC) Transfusion Independent for at Least 182 Days
Description: For participants who became RBC transfusion independent for at least 182 days during the double-blind study period, the mean maximum change from baseline in hemoglobin is summarized.
Time Frame: Baseline, up to 52 weeks
Population: The modified intent-to-treat (mITT) population included all participants with centrally-confirmed Low- or Int-1-risk MDS with del 5q[31] and documented RBC transfusion dependence who had received ≥ 1 dose of study drug. MITT participants who were transfusion independent for >= 182 study days are included.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg
Number analyzed (Participants) | 3 | 20 | 23
g/dL | 2.0 (0.61) | 5.5 (1.79) | 6.0 (1.97)

5. Secondary Outcome: Participants' Response in Platelet Counts as Defined by the International MDS Working Group (IWG 2000) During Double-blind Period
Description: The International MDS Working Group (IWG) defines a major platelet response for participants with a pre-treatment platelet count of <100,000/mm^3 as an absolute increase of ≥30,000/mm^3 whereas a minor response is defined as a ≥50% increase in platelet count with a net increase greater than 10,000/mm^3 but less than 30,000/mm^3.
Time Frame: up to 52 weeks
Population: The modified intent-to-treat (mITT) population included all participants with centrally-confirmed Low- or Int-1-risk MDS with del 5q[31] and documented RBC transfusion dependence who had received ≥ 1 dose of study drug. Additionally, the participant must have had a baseline platelet count of <100,000/mm^3 to be included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg
Number analyzed (Participants) | 3 | 6 | 4
Participants
  Major | 0 | 1 | 1
  Minor | 0 | 0 | 0
  None | 3 | 5 | 3

6. Secondary Outcome: Participants' Response in Absolute Neutrophil Counts as Defined by the International MDS Working Group (IWG 2000) During Double-blind Period
Description: A major neutrophil response is defined by the International MDS Working Group (IWG) criteria as at least a 100% increase, or an absolute increase of ≥500/mm^3 for participants with absolute neutrophil counts (ANC) of less than 1,500/mm^3 before therapy, whichever is greater. A minor response for such participants is defined as an ANC increase of at least 100%, but absolute increase <500/mm^3.
Time Frame: up to week 52
Population: The modified intent-to-treat (mITT) population included all participants with centrally-confirmed Low- or Int-1-risk MDS with del 5q[31] and documented RBC transfusion dependence who had received ≥ 1 dose of study drug. Additionally, the participant must have had a baseline absolute neutrophil counts (ANC) < 1,000/mm^3.
Measure: Number; unit: Participants
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg
Number analyzed (Participants) | 10 | 18 | 17
Participants
  Major | 1 | 3 | 2
  Minor | 0 | 0 | 1
  None | 9 | 15 | 14

7. Secondary Outcome: Participants' Response Based on Bone Marrow Samples by the International MDS Working Group (IWG 2000) During Double-blind Period
Description: The IWG criteria for bone marrow improvement: a complete remission is bone marrow sampling showing less than 5% myeloblasts with normal maturation of all cell lines, with no evidence for dysplasia. A partial remission is ≥ 50% decrease in blasts over pre-treatment. Bone marrow progression is a ≥ 50% increase in blasts that exceed the top range of the pretreatment percentile range: a) <5% blasts b) 5-10% blasts c) 10-20% blasts d) 20-30% blasts. For example, a participant with <5% blasts pretreatment with an on study blast increase of 50% which is now >5% showed bone marrow progression.
Time Frame: up to 52 weeks
Population: Intent to treat population. Participants represented in the treatment groups to which they were randomized. Placebo response is limited to the double-blind phase. There were 10 responders in the placebo group who achieved their response under lenalidomide treatment after crossover to open-label.
Measure: Number; unit: Participants
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg
Number analyzed (Participants) | 67 | 69 | 69
Participants
  Complete remission | 0 | 7 | 12
  Partial remission | 0 | 5 | 1
  Stable Disease | 37 | 35 | 33
  Progression | 3 | 4 | 3

8. Secondary Outcome: Participants Showing Cytogenetic Response by the International MDS Working Group (IWG 2000) During Double-blind Period as Evaluated by Central Review
Description: The IWG criteria for evaluating cytogenetic response require a minimum of 20 baseline and post-baseline analyzable metaphases using conventional cytogenetic techniques. A major cytogenetic response is defined as no detectable cytogenetic abnormality if preexisting abnormality was present whereas a minor response requires ≥50% reduction in abnormal metaphases. Progression could be concluded based on as few as 3 metaphases if there were additional abnormalities. The best response is represented.
Time Frame: up to 52 weeks
Population: Modified intent to treat population, which is defined as participants with centrally-confirmed Low- or Int-1-risk MDS with del 5q[31] and documented RBC transfusion dependence who had received ≥ 1 dose of study drug. Participants had to have had more than 1 post-baseline assessment in order to be evaluable for cytogenetic response.
Measure: Number; unit: Participants
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg
Number analyzed (Participants) | 41 | 37 | 40
Participants
  Major response | 0 | 5 | 10
  Minor response | 0 | 3 | 7
  Cytogenetic progression | 5 | 10 | 8
  Not evaluable/data not available | 10 | 10 | 1

9. Secondary Outcome: Participants Who Progressed to Acute Myeloid Leukemia (AML) During the Study
Description: Number of participants who progressed to acute myeloid leukemia during the study, summarized at three different timepoints: first 16 weeks of the double-blind study, week 52 of the double-blind study, and up to 36 months which includes the double-blind and open-label periods of the study. The counts are cumulative by timeframe.
Time Frame: up to 3 years
Population: Intent to treat population. Participants represented in the treatment groups to which they were randomized.
Measure: Number; unit: Participants
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg
Number analyzed (Participants) | 67 | 69 | 69
Participants
  Double-Blind (first 16 weeks) | 2 | 2 | 0
  Double-Blind (52 weeks) | 4 | 7 | 2
  Double-Blind + Open-Label | 21 | 16 | 15

10. Secondary Outcome: Kaplan Meier Estimates of Overall Survival by Randomized Group
Description: Kaplan Meier estimate for median length of survival for study participants as they were randomized at the start of the study.
Time Frame: up to 3 years
Population: Safety population: All randomized participants who received any Lenalidomide or placebo.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg
Number analyzed (Participants) | 67 | 69 | 69
Months | 42.4 [31.9 to NA] — The confidence interval cannot be estimated due to not enough number of deaths. | NA [24.6 to NA] — The confidence interval cannot be estimated due to not enough number of deaths. | 44.5 [35.5 to NA] — The confidence interval cannot be estimated due to not enough number of deaths.

11. Secondary Outcome: Participant Count of Deaths During Double-blind and Open-label by Randomized Group
Description: Count of participant deaths throughout the entire study and reported by the original treatment assignment.
Time Frame: up to 3 years
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg
Number analyzed (Participants) | 67 | 69 | 69
Participants | 35 | 32 | 34

12. Secondary Outcome: Change From Baseline in the Functional Assessment of Cancer Therapy-Anemia (FACT-An) Endpoints at Week 12
Description: The Functional Assessment of Cancer Therapy-Anemia (FACT-An) questionnaire (Yellen, 1997) was used to assess health-related quality of life (HRQoL).
  In addition to general HRQoL, the FACT-An measures the impact of fatigue and other anemia-related symptoms on patient functioning. The overall score range for the FACT-An is 0-188. Higher scores indicate better HRQoL.
Time Frame: Baseline, Week 12
Population: Participants who had both Baseline and Week 12 FACT-An data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg
Number analyzed (Participants) | 52 | 45 | 48
units on a scale | -2.5 (18.50) | 5.9 (18.26) | 5.8 (23.17)
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide 5 mg; Test type: Superiority or Other; p < 0.05, ANOVA
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide 10 mg; Test type: Superiority or Other; p < 0.05, ANOVA

13. Secondary Outcome: Change From Baseline in the Trial Outcome Index-Anemia (TOI-An) Endpoints at Week 12
Description: The Trial Outcome Index-Anemia (TOI-An) composed of the physical and functional subscales of the FACT-G along with the Anemia subscale was used to assess health-related quality of life (HRQoL). The overall score range for the TOI-An is 0-136. Higher scores indicate better HRQoL.
Time Frame: Baseline, Week 12
Population: Participants who had both Baseline and Week 12 TOI-An data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg
Number analyzed (Participants) | 52 | 46 | 49
units on a scale | -1.1 (17.13) | 5.6 (15.56) | 4.9 (18.16)
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide 5 mg; Test type: Superiority or Other; p = 0.054, ANOVA
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide 10 mg; Test type: Superiority or Other; p = 0.080, ANOVA

14. Secondary Outcome: Change From Baseline in the Trial Outcome Index-Fatigue (TOI-F) Endpoints at Week 12
Description: The Trial Outcome Index-Fatigue(TOI-F) composed of the physical and functional subscales of the FACT-G along with the fatigue items from the Anemia subscale was used to assess health-related quality of life (HRQoL). The overall score range for the TOI-F is 0-108. Higher scores indicate better HRQoL.
Time Frame: Baseline, Week 12
Population: Participants who had both Baseline and Week 12 TOI-F data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg
Number analyzed (Participants) | 53 | 46 | 49
units on a scale | -0.8 (14.76) | 4.8 (14.21) | 3.9 (15.47)
Statistical Analysis 1: Comparison: Placebo vs Lenalidomide 5 mg; Test type: Superiority or Other; p = 0.062, ANOVA
Statistical Analysis 2: Comparison: Placebo vs Lenalidomide 10 mg; Test type: Superiority or Other; p = 0.113, ANOVA

15. Secondary Outcome: Summary of Participants Who Had Adverse Events (AE) During the Double-blind Period
Description: Counts of study participants who had adverse events (AEs) during the double-blind period by MedDRA System Organ Class (SOC) and preferred term. A participant with multiple occurrences of an adverse event within a category is counted only once in that category. Adverse events were evaluated by the investigator.
  The National Cancer Institute (NCI)'s Common Terminology Criteria for AEs (CTCAE) was used to grade AE severity. Severity grade 3= severe and undesirable AE. Severity grade 4= life-threatening or disabling AE.
Time Frame: up to week 52
Population: Safety population.
Measure: Number; unit: participants
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg
Number analyzed (Participants) | 67 | 69 | 69
participants
  At least one AE | 64 | 69 | 69
  At least one AE related to study drug | 34 | 68 | 66
  At least one NCI CTCAE grade 3-4 AE | 29 | 62 | 65
  At least one related NCI CTCAE grade 3-4 AE | 13 | 61 | 61
  At least one serious AE | 14 | 31 | 32
  At least one serious AE related to study drug | 1 | 17 | 13
  An AE leading to discontinuation of study drug | 3 | 12 | 6
  An AE leading to dose reduction or interruption | 5 | 44 | 51
  Deaths within 30 days of last dose of study drug | 4 | 2 | 4

ADVERSE EVENTS:
Time Frame: Placebo arm is limited to the double-blind period. Lenalidomide 5 mg and 10 mg treatment arms cover both double-blind and open-label periods. The Placebo Crossover to 5 mg Open-label Period arm is limited to the open-label period.
Arm/Group | Placebo | Lenalidomide 5 mg | Lenalidomide 10 mg | Placebo Crossover to 5 mg Open-label Period
Serious Adverse Events (participants affected / at risk) | 14/67 | 42/69 | 42/69 | 33/56
Other Adverse Events (participants affected / at risk) | 64/67 | 69/69 | 69/69 | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=67) | Lenalidomide 5 mg (N=69) | Lenalidomide 10 mg (N=69) | Placebo Crossover to 5 mg Open-label Period (N=56)
Pyrexia (General disorders) | 2 | 5 | 2 | 3
Asthenia (General disorders) | 1 | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0
General Physical Health Deterioration (General disorders) | 0 | 0 | 2 | 0
Generalised Oedema (General disorders) | 0 | 1 | 0 | 0
Mucosal Inflammation (General disorders) | 0 | 0 | 1 | 0
Multi-Organ Failure (General disorders) | 0 | 0 | 0 | 1
Non-cardiac Chest Pain (General disorders) | 0 | 1 | 0 | 0
Arthritis Bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 5 | 3 | 1
Anal Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 1 | 0
Febrile Infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0
Neutropenic Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia Legionella (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0
Septic Shock (Infections and infestations) | 0 | 0 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 3 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0
Acute Respiratory Distress Syndrome (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 8 | 8 | 5
Acute Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Histiocytosis Haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Refractory Anaemia with an excess of blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 1
Cotard's Syndrome (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Mood Altered (Psychiatric disorders) | 0 | 1 | 1 | 0
Atrial Flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 2 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 2 | 0 | 2
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 2 | 1 | 3
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 1
Food Poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intussusception (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tooth Disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Meniscus Lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Synovial Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Transfusion Reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1 | 0
Coma (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 0
Urethral caruncle (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 1 | 0
Stress Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 1 | 4 | 3
Arterial Occlusive Disease (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Thrombophlebitis Superficial (Vascular disorders) | 0 | 0 | 0 | 1
Venous Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 4 | 1 | 1
Amaemia Haemolytic Autoimmune (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Autoimmune Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Bone Marrow Failure (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 3
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 5 | 5 | 5
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 6 | 3 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
International normalised Ratio Increased (Investigations) | 0 | 1 | 0 | 0
Urine Human Chorionic Gonadotropin Abnormal (Investigations) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Pyoderma Gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Cytogenetic Abnormality (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=67) | Lenalidomide 5 mg (N=69) | Lenalidomide 10 mg (N=69) | Placebo Crossover to 5 mg Open-label Period (N=56)
Diarrhoea (Gastrointestinal disorders) | 12 | 32 | 37 | 26
Nausea (Gastrointestinal disorders) | 6 | 16 | 21 | 11
Constipation (Gastrointestinal disorders) | 5 | 18 | 19 | 17
Abdominal Pain (Gastrointestinal disorders) | 4 | 7 | 14 | 10
Vomiting (Gastrointestinal disorders) | 4 | 8 | 9 | 3
Dry Mouth (Gastrointestinal disorders) | 2 | 4 | 5 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 8 | 8 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 4 | 5 | 4
Flatulence (Gastrointestinal disorders) | 0 | 2 | 1 | 4
Asthenia (General disorders) | 10 | 10 | 10 | 9
Fatigue (General disorders) | 5 | 17 | 17 | 11
Oedema Peripheral (General disorders) | 5 | 15 | 13 | 10
Chest Pain (General disorders) | 4 | 1 | 0 | 1
Pyrexia (General disorders) | 3 | 11 | 16 | 9
Non-Cardiac Chest Pain (General disorders) | 1 | 5 | 1 | 2
Influenza Like Illness (General disorders) | 0 | 5 | 5 | 1
Oedema (General disorders) | 0 | 3 | 4 | 1
Pain (General disorders) | 0 | 1 | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 12 | 55 | 57 | 45
Anaemia (Blood and lymphatic system disorders) | 6 | 10 | 6 | 13
Leukopenia (Blood and lymphatic system disorders) | 3 | 12 | 8 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 38 | 36 | 26
Nasopharyngitis (Infections and infestations) | 5 | 15 | 16 | 8
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 11 | 12 | 8
Urinary Tract Infection (Infections and infestations) | 4 | 6 | 12 | 8
Bronchitis (Infections and infestations) | 3 | 7 | 14 | 8
Cystitis (Infections and infestations) | 1 | 2 | 4 | 4
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 2 | 5 | 2
Respiratory Tract Infection (Infections and infestations) | 1 | 9 | 3 | 6
Sinusitis (Infections and infestations) | 1 | 1 | 6 | 4
Gastroenteritis (Infections and infestations) | 0 | 7 | 6 | 2
Gastroenteritis Viral (Infections and infestations) | 0 | 4 | 0 | 0
Influenza (Infections and infestations) | 0 | 5 | 5 | 3
Oral Herpes (Infections and infestations) | 0 | 6 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 3 | 4 | 0
Rhinitis (Infections and infestations) | 0 | 4 | 3 | 4
Headache (Nervous system disorders) | 6 | 12 | 14 | 5
Dizziness (Nervous system disorders) | 3 | 8 | 10 | 8
Paraesthesia (Nervous system disorders) | 3 | 8 | 3 | 6
Sciatica (Nervous system disorders) | 2 | 2 | 4 | 0
Balance Disorder (Nervous system disorders) | 0 | 0 | 4 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 4 | 1 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 6 | 12 | 15 | 13
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 12 | 8 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 6 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 6 | 5 | 5
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 5 | 10 | 9
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 8 | 8 | 8
Iron Overload (Metabolism and nutrition disorders) | 2 | 4 | 5 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 4 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 7 | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3 | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 12 | 10 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 12 | 9 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 4 | 3
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 3 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 6 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 16 | 20 | 7
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 10 | 10 | 6
Rash (Skin and subcutaneous tissue disorders) | 1 | 18 | 12 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 4 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 3 | 4 | 3
Insomnia (Psychiatric disorders) | 5 | 6 | 9 | 6
Depression (Psychiatric disorders) | 3 | 4 | 2 | 2
Anxiety (Psychiatric disorders) | 2 | 3 | 5 | 4
Contusion (Injury, poisoning and procedural complications) | 1 | 3 | 4 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 4 | 2
Joint Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 3
Wound (Injury, poisoning and procedural complications) | 0 | 2 | 4 | 1
Alanine Aminotransferase Increased (Investigations) | 2 | 7 | 5 | 4
Weight Decreased (Investigations) | 1 | 6 | 5 | 12
Atrial Fibrillation (Cardiac disorders) | 2 | 0 | 1 | 4
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 4
Haematoma (Vascular disorders) | 2 | 6 | 6 | 5
Phlebitis (Vascular disorders) | 1 | 1 | 4 | 2
Hypertension (Vascular disorders) | 0 | 7 | 9 | 5
Cataract (Eye disorders) | 0 | 1 | 5 | 2
Conjunctivitis (Eye disorders) | 0 | 0 | 5 | 2
Dysuria (Renal and urinary disorders) | 2 | 1 | 3 | 3
Vertigo (Ear and labyrinth disorders) | 1 | 8 | 3 | 2
Pneumonia (Infections and infestations) | 2 | 2 | 2 | 5
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 11 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Multicenter publication must include input from investigators and Celgene, agreement to be established before publication. It has priority over subset (single center) publication, for duration of 1 year after study completion.
* Individual investigators have publication right after multicenter publication is complete (or 1 year after study completion), whichever is first. In this case, Celgene has the right to comment and right to ask delay of publication for 90 days.